CLINICAL TRIAL: NCT02326454
Title: A Phase 2 Randomised, Double-blind, Placebo Controlled, Study of MR901 in Patients With Moderate to Severe Lower Urinary Tract Symptoms (LUTS) Due to Benign Prostatic Hyperplasia (BPH)
Brief Title: A Placebo Controlled Study of MR901 (Talaporfin Sodium Sodium + a Drug-activating Device) for the Relief of Lower Urinary Tract Symptoms Due to Benign Prostatic Hyperplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Light Sciences Oncology (Industry)
Collaborators: Mundipharma Research Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MR901-2501
Record Dates: First submitted 2014-12-16; First posted 2014-12-29 (Estimated); Last update posted 2018-08-08 (Actual); Status verified 2018-08

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia | interventions — Talaporfin; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Talaporfin sodium/Light dose 100 J/cm (Active Comparator): Single 1 mg/kg dose of talaporfin sodium is administered intravenously with Drug Activator 100 J/cm delivering light for 60 minutes of the 2-hour treatment period
  Interventions: Drug: talaporfin sodium; Device: Drug Activator 100 J/cm
- Talaporfin sodium/Light dose 200 J/cm (Active Comparator): Single 1 mg/kg dose of talaporfin sodium is administered intravenously with Drug Activator 200 J/cm delivering light for 2 hours
  Interventions: Drug: talaporfin sodium; Device: Drug Activator 200 J/cm
- Saline/Light dose 100 J/cm (Placebo Comparator): 0.9% Sodium Chloride is administered intravenously with Drug Activator 100 J/cm delivering light for 60 minutes of the 2-hour treatment period
  Interventions: Drug: Saline; Device: Drug Activator 100 J/cm
- Saline/Light dose 200 J/cm (Placebo Comparator): 0.9% Sodium Chloride is administered intravenously with Drug Activator 200 J/cm delivering light for 2 hours.
  Interventions: Drug: Saline; Device: Drug Activator 200 J/cm

INTERVENTIONS:
Drug: talaporfin sodium — 1 mg/kg
  Other Names: LS11; NPe6; mono-(L)-aspartyl chlorin e6; ME2906; Laserphyrin; MR901is the combination of talaporfin sodium and the drug-activating device
  Arms: Talaporfin sodium/Light dose 100 J/cm; Talaporfin sodium/Light dose 200 J/cm
Drug: Saline
  Other Names: Placebo
  Arms: Saline/Light dose 100 J/cm; Saline/Light dose 200 J/cm
Device: Drug Activator 100 J/cm — Light Dose: 100 J/cm
  Other Names: Litx™ BPH Device
  Arms: Saline/Light dose 100 J/cm; Talaporfin sodium/Light dose 100 J/cm
Device: Drug Activator 200 J/cm — Light Dose: 200 J/cm
  Other Names: Litx™ BPH Device
  Arms: Saline/Light dose 200 J/cm; Talaporfin sodium/Light dose 200 J/cm

SUMMARY:
This study investigates the safety and efficacy of a photosensitive drug (talaporfin sodium) activated by an intraurethrally placed drug-activating device. MR901 is a code used to identify the combination of talaporfin sodium and the drug-activating device. Two different light doses will be tested against placebo groups in this 4-arm study.

DETAILED DESCRIPTION:
At least 192 patients with moderate-to-severe LUTS caused by BPH will be randomized in a 2:2:1:1 ratio to receive a single treatment of talaporfin sodium activated by light at one of two light doses or placebo (saline) with light at either dose. Follow-up is planned for 52 weeks from the day of treatment, with assessment at 12 weeks for change in International Prostate Symptom Score and continued follow-up during the remaining 40 weeks to assess duration of effect, need for any intervention, and longer-term safety.

ELIGIBILITY:
Inclusion criteria:

1. Males aged ≥40 years, weighing ≤200 Kg and able to provide written, informed consent.
2. Documented symptoms of BPH-LUTS for 6 months or more.
3. For patients regularly taking their prescribed BPH medication, dose should have been stable for at least 6 months for 5-alpha reductase inhibitors and 3 months for other BPH medications.
4. For patients who have withdrawn from regularly taking their prescribed BPH medication, there should have been a 6 month washout period for 5-alpha reductase inhibitors and 3 months for other BPH medications.
5. Have a total International Prostate Symptom Score (IPSS; Qs 1-7) of ≥ 15 at both V1 and V2 with a difference between those visits of ≤ 4 points.
6. Prostate volume of 30 - 80 mL (inclusive).
7. Maximum urinary flow rate (Qmax): 5 - 15 mL/sec (assessed on two voids each of ≥ 150mL).
8. Prostate-specific antigen (PSA) ≤10 ng/mL.
9. Post-void residual (PVR) volume ≤200 mL measured by a urinary catheter or bladder ultrasound according to local standard practice.
10. Prostatic urethral length (PUL) of between 30 - 55mm (inclusive) as measured by TRUS.
11. Willing and able to comply with photosensitivity precautions

Exclusion criteria

1. Any minimally invasive or surgical treatment within the last 12 months, and is not currently undergoing intraprostatic injections for BPH or any other prostatic condition. In any case, all enrolled subjects must have, at Baseline cystoscopy, an appearance/presentation of the prostate that is consistent with BPH and compatible with possible response to the study test treatment.
2. Subjects weighing >200 Kg.
3. Subjects with a history or current evidence of any of the following:

   1. A bladder disease or condition co-exists, such as idiopathic over-active bladder (OAB) and is evaluated by the Investigator as the predominant etiology for the subject's voiding symptomatology. A score of 4 points or greater on the 3 item OAB Awareness Tool (OABV3) or a high rate of urinary frequency (>13xday and/or 4x/night) would require investigator specific evaluation in ascribing these symptoms to a bladder condition as opposed to lower urinary tract obstruction. i) If the former is the assessment, then the subject requires exclusion from the study. ii) If the latter is the assessment, then the subject may be deemed eligible for inclusion.

      The subject eligibility explanation must be captured in the patient source documents.
   2. Active urinary tract infection i.e. must have a screening urinalysis without signs of infection or negative urine culture. Must not have had a previous symptomatic urinary tract infection within 4 weeks of the study.
   3. Urethral stricture or any other anatomical feature that would complicate catheterisation.
   4. Interstitial cystitis.
   5. Predominant prostate middle lobe, as determined by the Investigator.
   6. Prostate or bladder cancer or bladder carcinoma-in-situ - in particular, evidence from digital rectal exam (DRE) of prostate abnormalities suggestive of cancer in the last 12 months.
   7. Any other absolute indication for urosurgical intervention (such as acute or frequent retention, currently untreated bladder or urethral stones, urethral strictures/bladder neck contracture (BNC)).
   8. Damage to the bladder neck which could interfere with study procedures.
4. PSA level in excess of >10 ng/ml. If the PSA measurement is 2.5-10 ng/ml and/or has shown a clinically significant concerning increase in the last 6 months, local standard of care must be pursued to ensure the possibility of prostate cancer has been followed up and ruled out prior to study entry.
5. Subjects who had had a prostate biopsy within 6 weeks prior to Screening.
6. Any neurological condition affecting the bladder or a history of a neurogenic or chronically decompensated bladder i.e. neurogenic bladder, Parkinson's disease, history of chronic prostatitis within the last 5 years.
7. Prior treatment for urinary incontinence.
8. Requirements for daily incontinence pads or devices.
9. Subjects in whom nocturia is due to etiologies other than their BPH-LUTS, such as neurogenic bladder, diabetic neuropathy, neurocongestive heart failure, hepatic failure, nephritic syndrome, sleep disorder.
10. Previous or concurrent clinically relevant cardiovascular or cerebrovascular disorder within 24 weeks prior to the study i.e. unstable angina pectoris, myocardial infarction, transient ischemic attack, or cerebrovascular accident (stroke) within the past 6 months, or peripheral arterial disease with intermittent claudication or Leriche's syndrome.
11. Presence of serious hepatic diseases, renal diseases, immunological diseases, or pulmonary diseases that are clinically relevant.
12. Unwilling to use contraception for 3 months following administration of study medication or with an interest in future fertility.
13. A prolonged QTcF interval at baseline and/or who are currently taking medication that prolongs QT interval ("prolonged QTcF interval" defined as > 450 ms).
14. Known sensitivity to porphyrin-type drugs or known history of porphyria.
15. Any contraindications to use of the study treatment.
16. Active alcohol or drug abuse.
17. Subject has clinical laboratory test results outside the reference ranges of the testing laboratory that are deemed to be clinically significant. Subjects with isolated test results that are outside the specified ranges and that are assessed as clinically insignificant will be allowed at the discretion of the Investigator, after discussion with the Sponsor's Medical Monitor/Study Physician, if appropriate. If a subject has 1 isolated test result outside the specific range that is deemed potentially clinically significant, rescreening may be allowed at the discretion of the Investigator, after discussion with the Medical Monitor/Study Physician
18. Subjects with known disorders of coagulation, apart from those receiving anticoagulant / antithrombotic / antiplatelet therapy in whom the dose of such medication must have been stable for at least 1 month prior to randomisation. In those receiving Vitamin K antagonists (warfarin, acenocoumarol, phenindione, etc) the INR value at baseline should be <3.0.
19. Inability or unwillingness to comply with the required photosensitivity precautions during the three weeks following study treatment.
20. Subjects taking medications with a recognised propensity for causing photosensitivity (such as amiodarone, tetracyclines, sulphonamides) that cannot be discontinued for the initial study period, namely from 14 days prior to administration of study medication until 28 days afterwards.
21. Subjects with medical or investigation results deemed unfit for study treatment, as determined by medical history, clinical laboratory tests, ECG results, and physical examination that, in the Investigator's opinion, preclude entry into the study.
22. Subjects who have received an investigational medicinal product within 30 days or 5 half-lives of the investigational product prior to study entry (defined as the start of the Screening Period).
23. Subjects who are incapable of giving informed consent or complying with the protocol.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 225 (Actual)
Dates: Start 2014-11; Primary Completion 2017-03-29 (Actual); Study Completion 2017-03-29 (Actual)

PRIMARY OUTCOMES:
International Prostate Symptoms Score (IPSS) Questionnaire | 12 weeks
  Change from baseline in the total International Prostate Symptom Score (IPSS, Questions 1-7)

SECONDARY OUTCOMES:
Modified International Prostate Symptoms Score (IPSS) Questionnaire | 1, 2 and 3 Weeks
  Modified IPSS used to evaluate subject's average experience of symptoms over preceding 7 days.
Patient Global Impression of Improvement (PGI-1) | 4, 12, 26 and 52 weeks
  The number of subjects in each of the 7 response categories will be collected by subject interview at all relevant time points
Clinical Global Impression of Improvement (CGI-1) | 4, 12, 26 and 52 weeks
  The number of subjects in each of the 7 response categories will be assessed by the Investigator at all relevant time points.
Maximum Urinary Flow Rate (Qmax) | 1, 2, 3, 4, 12, 26 and 52 weeks
  The maximum rate at which urine can be voided, as measured using free uroflowmetry using two measurement 'runs' on two separate voids of at least 150mL each (where possible).
Post-void residual volume (PVR volume) | 1, 2, 3, 4, 12, 26 and 52 weeks
  Measured post-voiding through insertion of a urinary catheter to complete bladder emptying, or measured by bladder ultrasound according to local standard practice.
3-Day Frequency/Volume Data | 1, 2, 3, 4, 12, 26 and 52 weeks
  Data on urinary frequency and void volume will be collected by subjects for 3 days prior to each clinic visit
Safety and tolerability assessed by the number of subjects with Adverse Events | 52 weeks
  Assessed by variables such as AEs, laboratory parameters, vital signs, ECGs
Prostate-specific Antigen (PSA) | 1, 2, 3, 4, 12, 26 and 52 weeks
  As measured in serum, to detect any changes that may be caused by the effects of the therapeutic intervention under study on prostatic tissue.
Duration of effect/time to next treatment and treatment selected | 52 weeks
  Subjects whose condition progresses such that an additional intervention is required during the 12-month study period may provide secondary evidence of efficacy, dependent upon their treatment allocation.
International Index of Erectile Function-15 (IIEF-15) | 4, 12, 26 and 52 weeks
  15-item, 5 domain scale collected by subject interview, relating to the subjects' experience of erectile function (and other sexual parameters) over the previous 4 weeks).
Quality of Life evaluation - Bother Score | 1, 2, 3, 4, 12, 26 and 52 weeks
  Question 8 of the IPSS (also known as the Bother Score), which asks the subject to state how he would feel if he had to spend the rest of his life with his urinary condition just the way it is now, according to a 7-point scale (from 0 = 'delighted' to 6 = 'terrible').
Over-active Bladder-V3 (OAB-V3) | 1, 2, 3, 4, 12, 26 and 52 weeks
  OAB symptoms will be assessed, by subject interview, using the 3-item OAB Awareness Tool (OAB-V3), under which the subject reports how much they have been bothered by 3 symptoms of OAB (without a specified time period) according to a 6-point scale ranging from 0 (not at all) to 5 (a very great deal) (maximum score, 15).
International Prostate Symptoms Score (IPSS) Questionnaire | 4, 26 and 52 weeks
  IPSS Total Score as Change from Baseline
IPSS Subscores. | 1, 2, 3, 4, 12, 26 and 52 weeks
  The changes from baseline for each of the 7 IPSS questions, as well as the totals for each of the 2 categories of symptoms - voiding symptoms (incomplete emptying, intermittency, weak stream, straining) and storage symptoms (frequency, urgency and nocturia).
Prostate volume | Baseline and 12 weeks
  As measured on TRUS, to detect any changes that may be caused by the effects of the therapeutic intervention under study on prostatic volume.
Quality of Life evaluation - BPH Impact Index (BPHII) | 4, 12, 26 and 52 weeks
  The BPHII asks the subject to assess the impact of four aspects of their urinary condition over the previous 4 weeks, according to a 4-point (questions 1 - 3) or 5-point scale (question 4) (maximum score, 13).

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Koch-Hulle — LSO
Locations (40):
- United States (40):
  - Anniston, Alabama
  - Huntsville, Alabama
  - Anchorage, Alaska
  - Laguna Hills, California
  - Los Angeles, California
  - Murrieta, California
  - San Diego, California
  - Tarzana, California
  - Denver, Colorado
  - Aventura, Florida
  - Bradenton, Florida
  - Coral Gables, Florida
  - Pompano Beach, Florida
  - St. Petersburg, Florida
  - Tampa, Florida
  - Bloomington, Indiana
  - Greenwood, Indiana
  - New Orleans, Louisiana
  - Greenbelt, Maryland
  - Towson, Maryland
  - Chestnut Hill, Massachusetts
  - Las Vegas, Nevada
  - Edison, New Jersey
  - Albuquerque, New Mexico
  - Garden City, New York
  - New York, New York
  - Newburgh, New York
  - Poughkeepsie, New York
  - Concord, North Carolina
  - Cincinnati, Ohio
  - Middleburg Heights, Ohio
  - Springfield, Oregon
  - Bala-Cynwyd, Pennsylvania
  - Bryn Mawr, Pennsylvania
  - Myrtle Beach, South Carolina
  - Knoxville, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Salt Lake City, Utah
  - Mountlake Terrace, Washington

FDAAA 801 VIOLATIONS:
- Issues in Letter Addressed Confirmed — The responsible party has responded, and this matter was resolved administratively. — issued 2023-11-22, released 2023-08-02, posted 2023-12-07
- Violation Identified — Failure to Submit — issued 2023-07-19, released 2018-08-06, posted 2023-07-31